CLINICAL TRIAL: NCT00619073
Title: PACT (Platelet Activity After Clopidogrel Termination)
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Sanofi (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CPFS 2008-1
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-04

CONDITIONS: Blood Platelets; Clopidogrel
Keywords: blood platelets; platelet aggregation inhibitors; antiplatelet drugs; clopidogrel
MeSH Terms: interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel + aspirin (Active Comparator): The subjects will be randomized to clopidogrel 75 mg plus aspirin 81 mg orally daily for 14 days. The study drug (i.e., clopidogrel) will then be discontinued and aspirin continued for another 43 days.
  Interventions: Drug: clopidogrel + aspirin; Drug: Aspirin
- Placebo + aspirin (Placebo Comparator): The subjects will be randomized to placebo plus aspirin 81 mg orally daily for 14 days. The study drug (i.e., placebo) will then be discontinued and aspirin continued for another 43 days.
  Interventions: Drug: placebo; Drug: Aspirin

INTERVENTIONS:
Drug: clopidogrel + aspirin — Clopidogrel 75mg plus aspirin 81mg, tablet by mouth daily for 14 days.
  Other Names: Plavix; aspirin
  Arms: Clopidogrel + aspirin
Drug: placebo — Placebo plus aspirin 81 mg, tablet by mouth daily for 14 days.
  Other Names: aspirin
  Arms: Placebo + aspirin
Drug: Aspirin — Aspirin 81mg tablet by mouth continued daily alone for 43 days after day 14.

SUMMARY:
Clopidogrel is a medication that is used to decrease the ability of platelets to form blood clots.

The theory has been proposed that, in patients with coronary artery disease or stroke, increased platelet function after discontinuation of clopidogrel therapy is associated with an increased clotting risk. However, this theory has never been rigorously tested.

The goal of this research is to determine whether discontinuation of clopidogrel results in increased platelet function.

DETAILED DESCRIPTION:
In this study, we will address the question: does discontinuation of clopidogrel result in platelet hyperreactivity? We will perform a double-blind, placebo-controlled, crossover study in normal subjects, in whom platelet reactivity will be measured before clopidogrel or placebo, during clopidogrel or placebo, and at various time points after discontinuation of clopidogrel or placebo. The dose of clopidogrel will be the standard, FDA-approved dose: 75 mg daily. All subjects will be treated with aspirin 81 mg daily throughout the 57 days of study assessment in both the clopidogrel arm and the placebo arm, because the clinically relevant question is: in patients who remain on aspirin, does discontinuation of clopidogrel result in platelet hyperreactivity?

ELIGIBILITY:
Inclusion Criteria:

* Must be a normal healthy subject
* Must be between 21-70 years old
* Must be able to take aspirin and clopidogrel.
* Must be able to have blood drawn 16 times over approximately 3 months.

Exclusion Criteria:

* Subject who is currently taking aspirin or another anti-platelet drug such as clopidogrel. Subject must be free of these medications for 10 days before enrolling in this study.
* Subject who is currently taking a non-steroidal anti-inflammatory drug such as ibuprofen or naproxen. Subject must be free of these medications for 3 days before enrolling in this study.
* Subject who is currently taking medications for depression or medications that lower blood pressure or lower blood sugar.
* Subject who are pregnant or may become pregnant during the study or who is breast feeding.
* Subject with a known allergy to aspirin or clopidogrel.
* Cigarette smoking or use of other nicotine product.
* Subject with a history of any of the following: coronary artery disease; stroke; bleeding disorder; ongoing bleeding; previous life-threatening hemorrhage; stomach ulcers; gastrointestinal bleeding within the past 1 month; major surgery within the past 1 month; minor surgery within the past 2 weeks; or platelet transfusion within the past 7 days.
* Subject with a blood count, measured on the pre-study drug blood sample, that is not in the normal range.
* Subject who is enrolled in another clinical trial of an investigational drug.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan D. Michelson, M.D., Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Frelinger AL 3rd, Barnard MR, Fox ML, Michelson AD. The Platelet Activity After Clopidogrel Termination (PACT) study. Circ Cardiovasc Interv. 2010 Oct;3(5):442-9. doi: 10.1161/CIRCINTERVENTIONS.110.937961. Epub 2010 Aug 24. PMID 20736449
- See also: Home page of the study principal investigator — http://www.platelets.org/director.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited at UMass Medical School in Worcester, MA between April 2008 and May 2009.
Pre-assignment Details: 15 healthy participants recruited; 16 screened, 1 excluded (1 did not meet inclusion criteria).
Groups:
- Clopidogrel Then Placebo: The subjects will be randomized to clopidogrel 75 mg plus aspirin 81 mg orally daily for 14 days. The study drug (i.e., clopidogrel) will then be discontinued and aspirin continued for another 45 days. After a 30 day washout from completion of first intervention, the subjects will be crossed over to placebo plus aspirin 81 mg orally daily for 14 days. The study drug (i.e. placebo) will then be discontinued and aspirin continued for another 45 days.
- Placebo Then Clopidogrel: The subjects will be randomized to placebo plus aspirin 81 mg orally daily for 14 days. The study drug (i.e., placebo) will then be discontinued and aspirin continued for another 45 days. After a 30 day washout from completion of first intervention, the subjects will be crossed over to clopidogrel 75 mg plus aspirin 81 mg orally daily for 14 days. The study drug (i.e. clopidogrel) will then be discontinued and aspirin continued for another 45 days.
Period: First Intervention - 60 Days
Arm/Group | Clopidogrel Then Placebo | Placebo Then Clopidogrel
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout Period (30 Days)
Arm/Group | Clopidogrel Then Placebo | Placebo Then Clopidogrel
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention - 60 Days
Arm/Group | Clopidogrel Then Placebo | Placebo Then Clopidogrel
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive clopidogrel + aspirin first and placebo + aspirin first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 15
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Platelet Surface Activated GPIIb-IIIa Complex at 45 Days After Intervention.
Description: Value at 45 days after intervention minus value at baseline in platelet surface activated GPIIb-IIIa complex using flow cytometry.The types and concentrations of agonists used in the flow cytometry assays reported here were: ADP 0.5, 1, and 20 µmol/L; thrombin receptor activating peptide (TRAP) 1 and 20 µmol/L; and a combination of collagen 5 µg/mL and epinephrine 5 µmol/L. Mean Florescence Intensity (MFI) is used as unit of measure. MFI indicates relative degree of shift in fluorescence intensity of a population of platelets in arbitrary units.
Time Frame: Baseline and 45 days after intervention
Measure: Mean (Standard Error); unit: mean fluorescence intensity (MFI)
Arm/Group | Clopidogrel + Aspirin | Placebo + Aspirin
Number analyzed (Participants) | 15 | 15
mean fluorescence intensity (MFI) | 123.2 (17.6) | 126.7 (17.9)

ADVERSE EVENTS:
Arm/Group | Clopidogrel + Aspirin | Placebo + Aspirin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No